CLINICAL TRIAL: NCT06975319
Title: A Prospective, Randomised, Placebo-controlled, Double-blind First in Human Trial Evaluating the Safety and Immunogenicity of V-212 Administered on Three Occasions in Healthy Adult Volunteers.
Brief Title: Phase I Study With V-212 Vaccinations in Healthy Adult Volunteers
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virometix (Industry)
Collaborators: CR2O (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VMX-SPN-212-001; 2024-516008-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Immunisation Against Streptococcus Pneumoniae
Keywords: Healthy volunteer; Dose-finding; Safety; Immunogenicity; Placebo; Vaccination

STUDY DESIGN:
Intervention Model Description: Subjects will be healthy adults (male and female) aged between 18 and 45 years inclusive. A total of 60 subjects will be enrolled. 45 subjects will be vaccinated with V-212, and 15 subjects will receive placebo. Each subject will receive a total of 3 intramuscular (IM) injections of V-212 vaccine or placebo.
  Within each cohort there will be two times sentinel dosing applied (two subjects receive a single dose of the active IMP V-212 and one subject receives placebo). The enrolment of the sentinel subjects in the three cohorts will commence once at least 48 hours safety data (Day 2) have been reviewed by the investigator (and/or delegate) before the remaining subjects in the cohort will be enrolled.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (LD) Cohort (Experimental): Low Dose (LD) Cohort with 20 subjects; 15 will be vaccinated with V-212 and 5 subjects with placebo.
  Interventions: Biological: V-212 (or Placebo) administered by i.m injection (3 vaccinations) - low dose
- Intermediate Dose (MD) Cohort (Experimental): Intermediate Dose (MD) Cohort with 20 subjects; 15 will be vaccinated with V-212 and 5 subjects with placebo.
  Interventions: Biological: V-212 (or Placebo) administered by i.m injection (3 vaccinations) - medium dose
- High Dose (HD) Cohort (Experimental): High Dose (HD) Cohort with 20 subjects; 15 will be vaccinated with V-212 and 5 subjects with placebo.
  Interventions: Biological: V-212 (or Placebo) administered by i.m injection (3 vaccinations) - high dose

INTERVENTIONS:
Biological: V-212 (or Placebo) administered by i.m injection (3 vaccinations) - low dose — V-212 is a peptide antigen-based vaccine.
  Arms: Low Dose (LD) Cohort
Biological: V-212 (or Placebo) administered by i.m injection (3 vaccinations) - medium dose — V-212 is a peptide antigen-based vaccine.
  Arms: Intermediate Dose (MD) Cohort
Biological: V-212 (or Placebo) administered by i.m injection (3 vaccinations) - high dose — V-212 is a peptide antigen-based vaccine.
  Arms: High Dose (HD) Cohort

SUMMARY:
Virometix AG, is conducting research into a vaccine (V-212) to prevent pneumococcal disease, which is any type of illness caused by infection with a bacterium called Streptococcus pneumoniae (S. pneumoniae).

This trial is being conducted to obtain insight into the body's immune response and possible adverse effects of the trial vaccine in healthy adult volunteers. Three different doses will be evaluated to identify an optimal dose for future trials.

The trial is a prospective (collects data into the future), randomised, double-blind, phase I, first in human, placebo-controlled trial which will be conducted at one centre in Belgium. A total of 60 trial participants will be enrolled.

DETAILED DESCRIPTION:
Streptococcus pneumoniae (Spn) is a leading cause of a wide range of serious bacterial infections including otitis media, pneumonia, meningitis, and bacteraemia, with considerable morbidity and mortality worldwide. Prophylaxis is based on capsular polysaccharide vaccines which currently cover up to 23 serotypes. With the emergence of serotypes that are not well covered by existing vaccines (e.g. Serotypes 3 and 19A) and the increasing prevalence of non-vaccine serotypes which cannot be sustainably addressed by current vaccination strategies, there is an urgent need for an enhanced serotype-independent S. pneumoniae vaccine. V-212 is a novel peptide antigen vaccine with the potential to elicit serotype-independent protective immunity against S. pneumoniae infection by targeting conserved peptide regions found in all bacterial serotypes. This trial will evaluate the safety and immunogenicity of V-212 in healthy adults. The data generated will help establish the potential for V-212 to be further developed for vaccination of vulnerable populations such as elderly, immunocompromised, and paediatric patients.

Primary trial objective:

• To assess the safety and reactogenicity of vaccination with V-212 administered three times at 3 different dose levels compared with placebo.

Secondary trial objective:

• To assess the immunogenicity of vaccination with V-212 administered three times at 3 different dose levels compared with placebo.

Exploratory trial objectives:

* To assess native epitope recognition by V-212 IgG
* To evaluate cellular immunity
* To evaluate B-cell memory responses

Subjects will be healthy adults (male and female) aged between 18 and 45 years inclusive. A total of 60 subjects will be enrolled. 45 subjects will be vaccinated with V-212, and 15 subjects will receive placebo. Each subject will receive a total of 3 intramuscular (i.m.) injections of V-212 vaccine or placebo.

Within each cohort there will be sentinel dosing applied (two subjects receive a single dose of the active IMP). The enrolment of the sentinel subjects in the three cohorts will commence once at least 48 hours safety data (Day 2) have been reviewed by the investigator (and/or delegate) before the remaining subjects in the cohort will be enrolled.

The duration of the trial for each subject will be approximately 14 months. The total duration of the trial will be approximately 20 months with 9 months planned for recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Written signed informed consent obtained before any trial-related activities.
2. Healthy male and females aged between 18-45 years inclusive.
3. No evidence of clinically significant disease based on medical his-tory, physical examination, vital signs (blood pressure, heart rate, body temperature), laboratory safety parameters and clinical judgement.
4. Capable of meeting and complying with the requirements of the trial.
5. Female subjects of childbearing potential should have a negative serum pregnancy test at screening and must agree to use highly effective and acceptable contraceptive measures (as per the HMA/CTFG recommendations) 60 days before trial entry and during the active phase of the trial up to 2 months after the last dose (Day 150). Contraceptive measures considered adequate are:

   1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
   2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
   3. intrauterine device (IUD)
   4. intrauterine hormone-releasing system ( IUS)
   5. bilateral tubal occlusion
   6. vasectomised partner
   7. sexual abstinence
6. Levels of baseline immunity

   1. Subjects demonstrating baseline levels of immunity against V-212 epitopes that correspond to an OD450 value of below 0.8, when the ELISA IgG determination assay is performed with a serum sample at a 1:300 dilution.
   2. Subjects demonstrating baseline levels of immunity against one epitope that correspond to an OD450 value of below 2.0, while at the same time baseline levels of immunity against a second epitope are below 0.8, when the ELISA IgG determination assay is similarly performed.
   3. Subjects demonstrating baseline levels of immunity against one epitope that correspond to an OD450 value of below 2.0, while at the same time baseline levels of immunity against a second epitope are below 0.8, when the ELISA IgG determination assay is similarly performed.
7. Subject agrees not to participate in another interventional trial while participating in the present trial.

Exclusion Criteria:

1. Subject has had previous vaccination with any licensed or investigational pneumococcal vaccine at any time.
2. Presence of any tattoos on the injection site which make evaluation of the injection site impossible.
3. Subject has a history of microbiologically-proven invasive disease caused by Streptococcus pneumoniae.
4. Presence of serologic markers of acute or chronic Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBsAG and anti-HBc) and Hepatitis C Virus (anti-HCV) infections(s).
5. Any chronic disease, or history of significant disease that might interfere with the trial's conduct or completion. Some conditions may be accepted if stabilised, e.g. hypertension, based on clinical judgement.
6. An uncontrolled or poorly controlled active respiratory disease requiring medication.
7. Administration of systemic immunosuppressant or immuno-modifying drugs within the three month period, prior to trial start.
8. Confirmed or suspected (at the discretion of the Investigator) immune-suppressive or immune-deficient condition.
9. Current smokers. Ex-smokers must have discontinued at least 1 year or more prior to trial start.
10. Blood transfusion, blood product, immunoglobulins, received during the period of 3 months prior to trial start.
11. Clinically significant (according to Investigator's judgement) out of range laboratory values (referring to the FDA Guidance for Toxicity Grading Scale for volunteers in vaccine trials). The ab-normal lab test can be neglected if its cause is evident and of no clinical relevance.
12. Acute disease and/or fever (≥38°C measured by the oral route) at the time of IMP administration. Vaccine administration can be postponed until the febrile episode is over.
13. Recent vaccination (e.g., vaccine administration within 2 weeks (inactivated) or 4 weeks (live attenuated)) before each vaccination or evidence that a vaccine will be required during the trial period (e.g., planned travel).
14. Pregnant or plan to become pregnant during the trial period.
15. Breastfeeding.
16. Any other significant finding including a history of serious reactions to vaccines, that would increase, according to the Investigator, the risk of having an adverse outcome from participating in the trial.
17. History of any reaction or hypersensitivity likely to be exacerbated by any component of the investigational vaccine.
18. Alcohol, prescription drug, or substance use/abuse that, in the opinion of the Investigator, might interfere with the trial conduct or completion.
19. Medical condition or use of medication(s) that can increase the risk of bleeding or haematoma from the blood sampling and intramuscular injection.
20. Subjects employed by the Sponsor, by the vendors working on behalf of the Sponsor, by the Investigator or the trial site, or close relatives of research staff working on this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
(Serious) adverse events | From enrollment to the end of treatment at month 4 (incl. subject diary data collection) and during follow-up until month 12.
  Number and percentage of subjects reporting (serious) adverse events and pregnancies. Incidence rates from the time of administration through 30 days post-administration, by treatment (vaccine/placebo) group and by cohort (dose). Descriptive analyses will be performed for the 7- and 30-day periods following each administration.
  (Serious) adverse events will be recorded in a subject diary incl. concomitant medication from enrollment until month 4. Causality and duration (start/stop date and time) will be recorded. SAEs (and pregnancies) will be followed up until month 12 and described using narratives.
  Intensity assessments will be based on FDA guideline for toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials incl. 4 severity levels: mild, moderate, severe, or potentially life threatening (grade 1 to 4).
Solicited local and systemic adverse events | During 7 days post-each administration
  Number and percentage of subjects reporting solicited local and systemic AEs reported in a subject diary. Incidence rates from the time of administration through 30 days post-administration, by treatment (vaccine/placebo) group and by cohort (dose). Descriptive analyses will be performed for the 7- and 30-day periods following each administration.
  Local solicited symptoms are pain, induration (cm) , erythema (cm) and swelling (cm). Systemic solicited symptoms are headache, fatigue, body temperature (measured orally in Celsius), generalised myalgia.
  Intensity assessments will be based on FDA guideline for toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials incl. 4 severity levels: mild, moderate, severe, or potentially life threatening (grade 1 to 4).
Laboratory safety parameters (hematology & biochemistry) | From enrollment to the end of treatment at month 4.
  Number and percentage of subjects presenting with safety laboratory abnormalities (hematology & biochemistry - in international units) considered clinically significant. Evaluated and presented in a descriptive way with comparisons made by treatment (vaccine/placebo) group and by cohort (dose) versus baseline.
  Intensity assessments will be based on FDA guideline for toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials incl. 4 severity levels: mild, moderate, severe, or potentially life threatening (grade 1 to 4).x
Vital signs | From enrollment to the end of treatment at month 4 and during follow-up until month 12.
  Number and percentage of subjects with vital sign modifications. Evaluated and presented in a descriptive way with comparisons made by treatment (vaccine/placebo) group and by cohort (dose) versus baseline.
  Vital sign measurements include: height (cm), weight (kg), oral temperature (Celsius), BMI (kg/m2), heart rate (bts/min), and blood pressure (mmHg). Oral body temperature will be assessed per subject eDiary during the 7 days after each administration.
  Intensity assessments will be based on FDA guideline for toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials incl. 4 severity levels: mild, moderate, severe, or potentially life threatening (grade 1 to 4).
Physical examination | From enrollment to the end of treatment at month 4 and during follow-up until month 12.
  Number and percentage of subjects with abnormalities detected at the time of physical examination. Evaluated and presentation in a descriptive way with comparisons made by treatment (vaccine/placebo) group and by cohort (dose) versus baseline.
  Intensity assessments will be based on FDA guideline for toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials incl. 4 severity levels: mild, moderate, severe, or potentially life threatening (grade 1 to 4).

SECONDARY OUTCOMES:
To assess the immunogenicity of vaccination with V-212 | From enrollment to the end of treatment at month 4 and at month 12.
  Determination of epitope specific levels of anti-V-212 antibodies using V-212 IgG ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Leroux-Roels, Professor, Dr., Principal Investigator — Center for Vaccinology (CEVAC), Ghent University Hospital
Locations (1):
- Center for Vaccinology (CEVAC), Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No